CLINICAL TRIAL: NCT06690424
Title: Clinical Studies of the Efficacy and Safety of Remimazolam for Anesthesia Induction and Maintenance in Elderly Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRCF-YXFN-202401029
Record Dates: First submitted 2024-11-05; First posted 2024-11-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-10

CONDITIONS: Efficacy and Safety
Keywords: remimazolam; anesthesia induction; continuous anesthesia
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The enrolled patients and the data collectors were blinded to the grouping status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group R (Experimental): This group is the experimental group with remimazolam for anesthesia induction and maintenance
  Interventions: Drug: Remimazolam
- group P (Active Comparator): This group is the control group with propofol for anesthesia induction and maintenance
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — remimazolam 0.2mg / kg was injected IV during the induction of anesthesia，and remimazolam 0.3-0.5mg / kg / h was administered IV during anesthesia maintenance.
  Other Names: R
  Arms: group R
Drug: Propofol — Propofol 1.5-2mg / kg was injected IV during the induction of anesthesia，and Propofol 2-3mg / kg / h was administered IV during anesthesia maintenance.
  Other Names: P
  Arms: group P

SUMMARY:
the investigators are conducting a clinical study on the efficacy and safety of remimazolam for induction and maintenance of anesthesia in elderly patients. Project number: CRCF-YXFN-202401029, funded by the Red Cross Foundation of China and will take more than 2 years to complete.

This is a single-center, randomized, controlled clinical study, randomized 60 elderly subjects undergoing general anesthesia for elective surgery. According to the random number method, propofol group (control group, group P) and remimazolam group (experimental group, group R), 30 cases in each group.

By participating in this study, it is possible to make anesthesia induction rapid and stable, stable intraoperative circulation, rapid recovery and safe and comfortable, reduce the Incidence of intraoperative awareness, arrhythmia, postoperative delusion, and so on, which is conducive to rapid postoperative recovery and reduce hospitalization costs.

DETAILED DESCRIPTION:
Research background: Rapid and steady anesthesia induction, stable intraoperative circulation, rapid recovery, safe and comfortable, and few adverse reactions are the goals of anesthesiologists. Accelerating the surgical turnover and improving the efficiency are the clinical problems that need to be solved. Clinical general anesthesia often adopts static inhalation compound anesthesia to give full play to the advantages of intravenous and inhalation anesthesia and reduce their respective adverse reactions. Remimazolam, as a new ultra-short-acting benzodiazepine sedative, is not widely used in elderly patients, but its rapid onset, short time half-life, less accumulation, little cardiopulmonary inhibition, no injection pain, and can be antagonized by flumazenil, showing an irreplaceable advantage.

Study objective: To observe the efficacy and safety of remimazolam for the induction and maintenance of anesthesia in elderly patients, and to provide a new option for anesthesia management in elderly and critically ill patients.

Study method: This topic adopts a single-center, prospective, randomized, controlled research method, and expects to include 60 elderly subjects with general endotracheal anesthesia for elective surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgery for clinically diagnosed thyroid tumors
2. Patients with general anesthesia
3. Patients requiring endotracheal intubation
4. American Society of Anesthesia gradeⅡ to grade Ⅲ
5. age 60-75 years old
6. body mass index was between 18 and 28
7. Patients or their family was clear about the study process and volunteered to participate.

Exclusion Criteria:

1. Patients with known allergy to remimazolam or with previous history of severe allergy and family history
2. Patients with long-term use of narcotic analgesics, sedatives, or non- steroidal anti-inflammatory drugs
3. Patients with drug taking, opioid dependence or tolerance
4. Patients with combined brain injury or intracranial hypertension
5. Patients with severe abnormal function of the heart, lung, liver, kidney and other major organs
6. Patients with bradycardia, with a heart rate lower than 55 beats / minute or a high atrioventricular block
7. Patients with a previous history of allergic disease
8. Patients with a previous history of mental illness
9. Patients with a foreseeable difficult airway
10. The investigator does not consider it appropriate to attend this clinical investigator.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of induction of anesthesia | At 5 minutes after the onset of anesthesia induction
  Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≤ 1 point within 5 minutes of administration (The rating scale ranges from levels 0 to 5, and lower MOAA / S score indicates deeper depth of sedation, namely a higher scores mean a worse outcome. )

SECONDARY OUTCOMES:
Supplement rate of the study drug | During the operation period
  Number of patients requiring remimazolam supplementation / total number of patients in the experimental group
Sedation depth | At the beginning of induction (T0); bispectral index at 60 (T1); at 1minute after endotracheal intubation (T2); at surgical skin incision (T3), 30 minutes after the start of surgery(T4), at the end of surgery (T5), and 1minute (T6) after extubation
  the Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score at the different time points (The rating scale ranges from levels 0 to 5, and lower MOAA / S score indicates deeper depth of sedation, namely a higher scores mean a worse outcome. )
Amount of sedative and analgesic drugs used | During anesthesia maintenance period
  Amount of sedation and analgesics used per unit time during anesthesia maintenance period
Hemodynamic index （1） | At the beginning of induction (T0); bispectral index at 60 (T1); at 1minute after endotracheal intubation (T2); at surgical skin incision (T3), 30 minutes after the start of surgery(T4), at the end of surgery (T5), and 1minute (T6) after extubation
  Heart rate
Hemodynamic index （2） | At the beginning of induction (T0); bispectral index at 60 (T1); at 1minute after endotracheal intubation (T2); at surgical skin incision (T3), 30 minutes after the start of surgery(T4), at the end of surgery (T5), and 1minute (T6) after extubation
  mean arterial pressure

OTHER OUTCOMES:
General data of the patient | Before the operation
  Gender, age, height, weight, current medical history, history of combined diseases and medication allergy, history of hypertension / diabetes (maximum hypertension / blood glucose, type and age of medication, and complications of other organs)
Perioperative adverse events | up to 24 hours after surgery
  Incidence of intraoperative awareness, arrhythmia, postoperative delusion, and so on
Patient satisfaction questionnaire | up to 24 hours after surgery
  The rating scale ranges from levels dissatisfaction, basic satisfaction, satisfaction to very satisfaction, the higher scores mean a better outcome.
Peri-operative-related indicators（1） | up to 6 hours after surgery
  Operation time
Peri-operative-related indicators（2） | up to 6 hours after surgery
  extubation time
Peri-operative-related indicators（3） | up to 6 hours after surgery
  Wake up time
Peri-operative-related indicators（4） | up to 12 hours after surgery
  residence time of Post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Xiao MB Director of scientific research Department, Doctor, Principal Investigator — The Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Affiliated Hospital, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No